CLINICAL TRIAL: NCT06194877
Title: A Phase 1b, Open-Label, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, and Antitumor Activity of BGB-3245 With Panitumumab in Patients With Advanced or Metastatic RAS Mutant Colorectal and Pancreatic Ductal Cancers
Brief Title: A Study to Investigate BGB-3245 (Brimarafenib) With Panitumumab in Participants With Advanced or Metastatic RAS Mutant Colorectal and Pancreatic Ductal Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding terminated due to business reasons
Sponsor: MapKure, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3245-EGFR-001
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Pancreatic Ductal Cancer; Advanced or Metastatic RAS Mutant Colorectal and Pancreatic Ductal Cancers
Keywords: Advanced or Metastatic RAS mutant Colorectal and Pancreatic Ductal Cancers; BGB-3245; Panitumumab; Brimarafenib; BRAF; KRAS; NRAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Finding Part (Experimental): Participants with advanced or metastatic CRC and with known mutation status and tumor harboring an oncogenic mutation of BRAF, KRAS, or NRAS and with documented disease progression by RECIST during or after at least 1 line of prior therapy will be enrolled into 4 planned sequentially run cohorts. Participants will receive escalating doses of BGB-3245 in combination with panitumumab to establish the MTD and RP2D by assessing the safety, tolerability, preliminary antitumor activity, and pharmacokinetics (PK) for the combination of BGB-3245 with panitumumab.
  Interventions: Drug: BGB-3245; Drug: Panitumumab
- Part 2: Dose Expansion Part, Group 1 (Experimental): Participants with advanced or metastatic CRC that harbors KRAS or NRAS mutations who have been treated and had documented disease progression by RECIST criteria during or after at least 1 line of prior therapy. Participants will receive the RP2D of BGB-3245 in combination with panitumumab to further evaluate the safety, PK, and assess the preliminary antitumor activity of the RP2D of the BGB-3245 and panitumumab combination.
  Interventions: Drug: BGB-3245; Drug: Panitumumab
- Part 2: Dose Expansion Part, Group 2 (Experimental): Participants with advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) that harbors KRAS mutations who have been treated and had documented disease progression by RECIST criteria during or after at least 1 line of prior therapy. Participants will receive the RP2D of BGB-3245 in combination with panitumumab to further evaluate the safety, PK, and assess the preliminary antitumor activity of the RP2D of the BGB-3245 and panitumumab combination.
  Interventions: Drug: BGB-3245; Drug: Panitumumab

INTERVENTIONS:
Drug: BGB-3245 — Oral capsule
  Other Names: Brimarafenib
Drug: Panitumumab — Intravenous (IV) infusion via an infusion pump
  Other Names: Vectibix®

SUMMARY:
The primary objectives of Part 1 of this study are to:

* Assess the safety and tolerability of the combination of BGB-3245 and panitumumab in participants with advanced or metastatic colorectal cancer (CRC) with a known mutation status and tumor harboring an oncogenic mutation of v-Raf murine sarcoma viral oncogene homolog B; B-RAF proto-oncogene, serine/threonine kinase (BRAF), Kirsten rat sarcoma viral oncogene homolog (KRAS), or neuroblastoma RAS viral oncogene homolog (NRAS) with documented disease progression during or after at least 1 line of prior therapy.
* Determine the maximum tolerated dose (MTD) of BGB-3245 in combination with panitumumab and the recommended phase 2 dose (RP2D) of the combination.

The primary objective of Part 2 of this study is to determine the objective response rate (ORR) as assessed by initial investigator review using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 with BGB-3245 and panitumumab combination treatment at the RP2D.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with histologically confirmed advanced or metastatic solid tumors who have had documented disease progression by RECIST criteria during or after at least 1 prior line of systemic anticancer therapies in the representative population or are unable to receive standard of care therapy(ies) as noted by local guidelines.
2. Part 1 (Dose Finding): Participants with CRC with a known mutation status by local testing and tumor harboring an oncogenic mutation of BRAF, KRAS, or NRAS in the archival tumor sample or fresh tumor biopsy.
3. Part 2 (Dose Expansion): Participants must have a known mutation status by local testing and meet one of the following criteria according to the group they are enrolled into: Group 1: Participants with CRC that harbors KRAS or NRAS mutations in the archival tumor sample or fresh tumor biopsy. Group 2: Participants with PDAC that harbors KRAS mutations in the archival tumor sample or fresh tumor biopsy.
4. Participants must provide archival tumor tissue or a fresh tumor biopsy for retrospective mutation status analysis.
5. Participants must have radiologically measurable disease as defined per RECIST v1.1 at screening.
6. Eastern Cooperative Oncology Group performance status of ≤1 at screening.
7. Adequate hematologic and organ function, as indicated by defined laboratory values, prior to Cycle 1 Day 1.
8. Adequate cardiac function.

Key Exclusion Criteria:

1. Participants receiving cancer therapy (chemotherapy or other systemic anticancer therapies, immunotherapy, radiation therapy, or surgery) at the time of Cycle 1 Day 1.
2. Active infection requiring systemic treatment at the start of the study treatment.
3. Clinically significant cardiovascular disease and / or events within 6 months of signing the informed consent form.
4. Participants with toxicities that have not recovered to Grade ≤1 or stabilized and those Grade 2 toxicities listed as permitted in other eligibility criteria.
5. Participants with a history of pneumonitis or interstitial lung disease.
6. Participants with immune-related toxicities that have not resolved with appropriate management.
7. History or presence of gastrointestinal disease or other condition known to interfere with the absorption of drugs.
8. History of ulcerative colitis or Crohn's disease or protracted and ongoing immune-mediated diarrhea from prior checkpoint inhibitor use.
9. History of corneal perforation, keratitis, or severe dry eye.
10. Current evidence of symptomatic central nervous system metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression.
11. Any active malignancy ≤3 years before Cycle 1 Day 1 except for the specific cancer under investigation in this study and any localized or noninvasive cancer that has been treated curatively.
12. Known hypersensitivity to rapidly accelerated fibrosarcoma (RAF) inhibitors, anti-epidermal growth factor receptor (EGFR) monoclonal antibodies, or their excipients.
13. Any known history of Grade ≥3 toxicity lasting >14 days from another RAF, mitogen activated protein kinase, extracellular signal-regulated kinase, or anti-EGFR antibody inhibitor requiring discontinuation of treatment from these drugs.
14. Receiving any treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducer ≤14 days (or 5 half-lives, whichever is longer) before Cycle 1 Day 1 and until completion of dosing with BGB-3245 for at least 5 half-lives.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply. Summary of key criteria provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Serious Adverse Events (SAEs) | Up to approximately 2 years
Part 1: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 2 years
Part 1: Number of Participants with Adverse Events of Special Interest (AESIs) | Up to approximately 2 years
Part 1: Number of Participants with Interruptions to Dosing with BGB-3245 | Up to approximately 2 years
Part 1: Number of Participants with Reductions in Dosing with BGB-3245 | Up to approximately 2 years
Part 1: MTD of BGB-3245 | Up to approximately 2 years
Part 1: RP2D of BGB-3245 | Up to approximately 2 years
Part 2: ORR as Assessed by Initial Investigator Review | Up to approximately 2 years

SECONDARY OUTCOMES:
Part 1 and 2: Plasma Concentrations of BGB-3245 and Any Relevant Metabolites | Day 1 of each 28 day cycle (up to approximately 2 years)
Part 1: ORR as Assessed by Investigator Review using RECIST v1.1 | Up to approximately 2 years
Part 2: ORR as Assessed by Central Review | Up to approximately 2 years
Part 1 and 2: Duration of Response (DoR) | Up to approximately 2 years
Part 1 and 2: Disease Control Rate (DCR) | Up to approximately 2 years
Part 1 and 2: Progression Free Survival (PFS) | Up to approximately 2 years
Part 2: Number of Participants with SAEs | Up to approximately 2 years
Part 2: Number of Participants with TEAEs | Up to approximately 2 years
Part 2: Number of Participants with AESIs | Up to approximately 2 years
Part 2: Number of Participants with Interruptions to Dosing with BGB-3245 | Up to approximately 2 years
Part 2: Number of Participants with Reductions in Dosing with BGB-3245 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - Duke Cancer Institute, Durham, North Carolina
  - USOR - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes